CLINICAL TRIAL: NCT02845375
Title: Effect of Neuromuscular Blockade and Reversal by Sugammadex Versus Neostigmine on Breathing When Hypoxic or Hypercapnic in Volunteers
Brief Title: Effect of Neuromuscular Blockade and Reversal on Breathing
Acronym: BREATH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Albert Dahan, Professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P16.025
Record Dates: First submitted 2016-07-14; First posted 2016-07-27 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Sugammadex; Neostigmine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PLACEBO (Placebo Comparator): Placebo (normal saline) will be administered following a period of muscle relaxation after which respiratory measurements will be obtained.
  Interventions: Drug: Placebo
- NEOSTIGMINE (Other): intravenous neostigmine will be administered following a period of muscle relaxation after which respiratory measurements will be obtained.
  Interventions: Drug: Neostigmine
- SUGAMMADEX (Experimental): intravenous sugammade will be administered following a period of muscle relaxation after which respiratory measurements will be obtained.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — Sugammadex will be administered following a period of muscle relaxation after wich respiratory measurements will be obtained.
  Arms: SUGAMMADEX
Drug: Neostigmine — Neostigmine will be administered following a period of muscle relaxation after wich respiratory measurements will be obtained.
  Other Names: NEO
  Arms: NEOSTIGMINE
Drug: Placebo — Placebo will be administered following a period of muscle relaxation after wich respiratory measurements will be obtained.
  Other Names: Normal saline
  Arms: PLACEBO

SUMMARY:
In this study the investigators will assess (i) the effect of partial neuromuscular blockade (NMB; TOF ratio 0.8 and 0.6) induced by low-dose rocuronium on the ventilatory response to isocapnic hypoxia and (ii) the effect over time (from TOF 0.6 to TOF 1.0) of the reversal by sugammadex, neostigmine or placebo in healthy volunteers.

Additionally the investigators will assess the effect of partial NMB (TOF ratio 0.6) induced by low-dose rocuronium on the ventilatory response to hypercapnia and effect over time (from TOF 0.6 to TOF 1.0) of the reversal by sugammadex, neostigmine or placebo in healthy volunteers.

DETAILED DESCRIPTION:
The carotid bodies, located at the bifurcation of the common carotid artery, play a crucial and life-saving role in the control of breathing in humans. The carotid bodies contain type 1 cells that are primarily sensitive to low oxygen concentrations in arterial blood. In response to low oxygen the carotid bodies send information to the brainstem respiratory centers and a brisk hyperventilatory response will be initiated ensuring an increase in uptake of oxygen via the lungs. Following surgery, a rapid return of the carotid body function is vital and persistent loss of carotid body function may result in respiratory complications that occur independent of the effects of anesthetics (incl. muscle relaxants) on respiratory muscles. Respiratory complications that are related to the loss of carotid body function include the inability to respond properly to hypoxia as well the inability to overcome upper airway obstruction. The latter is especially important in patients with sleep disordered-breathing and obese patients. These patients rely on the optimal function of their carotid bodies in response to hypoxia or upper airway closure.

Important neurotransmitters involved in the carotid body response to hypoxia include acetylcholine, which acts through local nicotinergic acetylcholine receptors. Apart from the observation that muscle relaxants (which are blockers of the acetylcholine receptors) affect the proper functioning of the carotid bodies, the investigators have no knowledge on the dynamic effects of muscle relaxants on carotid body function over time or on the relationship between carotid body function and Train-of-Four (TOF) ratio over time. Additionally, there is no data on the link between the use of NMB antagonists and return of carotid body function. Linking TOF ratio to carotid body function is of clinical importance as a possible relationship will allow clinicians to predict carotid body function from the TOF ratio. The latter is highly relevant as the investigators show in a previous trial that a large proportion of patients is extubated at TOF ratio's < 0.7.

Apart from the carotid bodies, chemoreceptors in the brainstem exist that are sensitive to hypercapnia. This response system is not under control of cholinergic neurotransmission. Since the investigators may assume that the hypercapnic ventilatory response is not influenced by muscle relaxants the investigators can use this response to calibrate the hypoxic ventilatory response as both responses are equally affected by the effect of muscle relaxants on muscle function.

As stated there is data on the effect of muscle relaxants on carotid body function at one fixed TOF ratio (TOF ratio fixed at 0.7). No data are available on:

1. Dynamic effect of carotid body function as measured by the hypoxic ventilatory response at TOF ratio's slowly changing from 0.6 to 1.0;
2. Dynamic effect of reversal of NMB by sugammadex versus neostigmine. Sugammadex and neostigmine are both reversal agents of neuromuscular blockade. At their institution the investigators use both agents in clinical practice but remain without knowledge on their effects on carotid body function. The current proposal is designed to study items 1 and 2 in healthy awake volunteers.

ELIGIBILITY:
Inclusion Criteria:

* male gender
* age 18 years and older
* body mass index < 30 kg/m2.

Exclusion Criteria:

* Known or suspected neuromuscular disorders impairing neuromuscular function;
* allergies to muscle relaxants, anesthetics or narcotics;
* a (family) history of malignant hyperthermia or any other muscle disease;
* any medical, neurological or psychiatric illness (including a history of anxiety).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will publish the paper. After publication the data are available
Time Frame: Mid 2019
Access Criteria: Request to the authors and approved protocol for data analysis to be submitted. A review committee will then decide wether the data will be shared, deepening on supplementary data analyses by the authors

REFERENCES:
- [Background] Eriksson LI, Sato M, Severinghaus JW. Effect of a vecuronium-induced partial neuromuscular block on hypoxic ventilatory response. Anesthesiology. 1993 Apr;78(4):693-9. doi: 10.1097/00000542-199304000-00012. PMID 8096684
- [Background] Eriksson LI, Lennmarken C, Wyon N, Johnson A. Attenuated ventilatory response to hypoxaemia at vecuronium-induced partial neuromuscular block. Acta Anaesthesiol Scand. 1992 Oct;36(7):710-5. doi: 10.1111/j.1399-6576.1992.tb03550.x. PMID 1359723
- [Background] Dahan A, Nieuwenhuijs D, Teppema L. Plasticity of central chemoreceptors: effect of bilateral carotid body resection on central CO2 sensitivity. PLoS Med. 2007 Jul 24;4(7):e239. doi: 10.1371/journal.pmed.0040239. PMID 17676946

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 46 subjects were enrolled.6 did not meet inclusion citeria. 40 subjects were randomized
Period: Overall Study
Arm/Group | PLACEBO | NEOSTIGMINE | SUGAMMADEX
Started | 13 | 14 | 13
Completed | 12 | 12 | 12
Not Completed | 1 | 2 | 1
Not completed — upper airway obstruction | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO | NEOSTIGMINE | SUGAMMADEX | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 12 | 36
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 20 [19 to 29] | 23 [18 to 29] | 23 [19 to 25] | 22 [18 to 29]
Sex: Female, Male [Count of Participants; unit: Participants] — All data were collectred during the screeing visit by an indpendent physician.
  Participants
    Sex: Female | 0 | 0 | 0 | 0
    Sex: Male | 12 | 12 | 12 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 12 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 12 | 12 | 12 | 36
Breathing response to a reduction in inspired oxygen concentration (hypoxic ventilatory response) [Mean (Standard Deviation); unit: L/min/% oxygen saturation] | 0.66 (0.21) | 0.43 (0.23) | 0.54 (0.16) | 0.55 (0.22)

OUTCOME MEASURES:

1. Primary Outcome: Breathing Increase Due to a Reduction in Inspired Oxygen Saturation (Hypoxic Ventilatory Response)
Description: The change in breathing response to a decrease in inspired oxygen concentration, which equals the isocapnic ventilatory response to hypoxia.
Time Frame: during the 1-2 hours following reversal
Population: Healthy male volunteers
Measure: Mean (Standard Deviation); unit: L/min/% desaturation
Arm/Group | PLACEBO | NEOSTIGMINE | SUGAMMADEX
Number analyzed (Participants) | 12 | 12 | 12
L/min/% desaturation
  Baseline | 0.66 (0.21) | 0.43 (0.22) | 0.54 (0.16)
  Relaxation | 0.34 (0.22) | 0.29 (0.22) | 0.31 (0.17)
  Reversal | 0.49 (0.13) | 0.36 (0.20) | 0.31 (0.17)

2. Primary Outcome: Breathing Increase Due to a Reduction in Inspired Oxygen Saturation (Hypoxic Ventilatory Response)
Description: The ventilatory response to a decrease in oxygen saturaytion of 80%
Time Frame: 0-10 minutes following reversal
Population: The ventilation-saturation data were analyzed using linear regreassion analysis. The slope is the acute hypoxic ventilatory response.
Measure: Mean (Standard Deviation); unit: L/min/%
Arm/Group | PLACEBO | NEOSTIGMINE | SUGAMMADEX
Number analyzed (Participants) | 12 | 12 | 12
L/min/% | 0.49 (0.13) | 0.36 (0.20) | 0.48 (0.13)
Statistical Analysis 1: Comparison: PLACEBO vs NEOSTIGMINE vs SUGAMMADEX; Test type: Superiority; p = 0.299, ANCOVA

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | PLACEBO | NEOSTIGMINE | SUGAMMADEX
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
There were no perceived limitations or caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-11-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT02845375/Prot_SAP_000.pdf
  • Informed Consent Form (2016-01-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT02845375/ICF_001.pdf